CLINICAL TRIAL: NCT03502694
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of Orally Administered Lumicitabine (JNJ-64041575) Regimens in Hospitalized Adult Subjects Infected With Human Metapneumovirus
Brief Title: Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of Oral Lumicitabine Regimens in Hospitalized Adult Participants Infected With Human Metapneumovirus
Acronym: STEP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108378; 2017-001696-22 (EudraCT Number); 64041575MPN2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Metapneumovirus
MeSH Terms: interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen A (Low-Dose Lumicitabine) (Experimental): Participants will receive a single 750 milligram (mg) loading dose (LD) (Dose 1) of lumicitabine and matching placebo followed by nine 250 mg tablets as maintenance doses (MDs) (Doses 2 to 10) of lumicitabine and matching placebo administered twice daily during Day 1 to Day 5/6 (depending on the timing of the LD).
  Interventions: Drug: Lumicitabine; Drug: Placebo
- Regimen B (High-Dose Lumicitabine) (Experimental): Participants will receive a single 1000 mg LD (Dose 1) of lumicitabine followed by nine 500 mg tablets as MDs (Doses 2 to 10) of lumicitabine and matching placebo tablet, administered twice daily during Day 1 to Day 5/6 (depending on the timing of the LD).
  Interventions: Drug: Lumicitabine; Drug: Placebo
- Regimen C (Placebo) (Placebo Comparator): Participants will receive a placebo LD (Dose 1) followed by nine MDs (Doses 2 to 10) of matching placebo, administered twice daily during Day 1 to Day 5/6 (depending on the timing of the LD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumicitabine — Participants will receive loading dose and maintenance dose of lumicitabine tablets orally.
  Other Names: JNJ-64041575, ALS-008176
  Arms: Regimen A (Low-Dose Lumicitabine); Regimen B (High-Dose Lumicitabine)
Drug: Placebo — Participants will receive matching placebo tablets orally.

SUMMARY:
The purpose of this study is to determine in hospitalized adult participants infected with human metapneumovirus (hMPV - a virus closely related to respiratory syncytial virus (RSV) and has been identified as an important cause of acute respiratory infections, affecting all age groups) the dose-response relationship of multiple regimens of lumicitabine on antiviral activity based on nasal hMPV shedding using quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR) assay.

DETAILED DESCRIPTION:
The study consists of 3 phases: screening phase, treatment phase (Day 1 to Day 5/6 [depending on timing of loading dose]), and follow-up phase of 28 days post randomization. Participants will have assessments at Days 7, 10, 14, and 28 to evaluate safety, efficacy, and pharmacokinetics (PK). The primary hypothesis of study is a positive dose-response relationship of active treatment on average hMPV viral load area under concentration versus time curve (AUC) over 7 days, meaning that either average AUC on pooled active treatments is lower than on placebo, or average AUC on high active dose is lower than average AUC on placebo using multiple contrast testing. Based on review of PK, efficacy and safety data, Independent Data Monitoring Committee (IDMC) may recommend modifications to study design that is changes in dose and treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Participants hospitalized (or in Emergency room prior to hospitalization) at the time of randomization and unlikely to be discharged for the first 24 hours after randomization
* Participants diagnosed with human metapneumovirus (hMPV) infection using a rapid polymerase chain reaction (PCR)-based molecular diagnostic assay, with or without coinfection with another respiratory pathogen (respiratory virus or bacteria)
* Participants with an acute respiratory illness with signs and symptoms consistent with a viral infection (for example, fever, cough, nasal congestion, runny nose, sore throat, myalgia, lethargy, shortness of breath, or wheezing) with onset less than or equal to (<=)5 days from the anticipated time of randomization
* With the exception of the symptoms related to hMPV infection, participants must be medically stable on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population, and/or the hMPV infection. This determination must be recorded in the participant's source documents and initialed by the investigator
* A woman must have a negative urine pregnancy test (beta-human chorionic gonadotropin [b-hCG]) at screening

Exclusion Criteria:

* Participants who are not expected to survive for more than 48 hours
* Participants who have had major thoracic or abdominal surgery in the 6 weeks prior to randomization
* Participants who are considered by the investigator to be immunocompromised within the past 12 months, whether due to underlying medical condition (for example, malignancy or genetic disorder) or medical therapy (for example, medications other than corticosteroids for the treatment of chronic obstructive pulmonary disease (COPD) or asthma exacerbations, chemotherapy, radiation, stem cell or solid organ transplant)
* Participants undergoing peritoneal dialysis, hemodialysis, or hemofiltration or with an estimated glomerular filtration rate (GFR, determined by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) of (<) 60 milliliters per minute (mL/min) per 1.73 meter square (m^2)
* Participants with a known history of human immunodeficiency virus (HIV) or chronic viral hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-05 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-10-28 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of Human Metapneumovirus (hMPV) Viral Load | Baseline up to Day 7
  The AUC of hMPV ribonucleic acid (RNA) logarithm base 10 (log10) viral load (measured by quantitative real time reverse transcriptase polymerase chain reaction [qRT-PCR] in the mid-turbinate nasal swab specimens) is estimated by analyzing mean log10 viral load values over time using a restricted maximum likelihood based repeated measures approach.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 28 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with an Abnormal Physical Examination Findings (Height, Body Weight, Respiratory System, Nose, Ear, Throat, Facial and Neck Lymph Nodes, and Skin Examination) as a Measure of Safety and Tolerability | Up to 28 days
  Number of participants with an abnormal physical examination will be reported. A complete physical examination (including all body systems, height [only at screening], and body weight measurement) or a directed physical examination including respiratory system, nose, ear, throat, facial and neck lymph nodes, and skin examination will be performed.
Number of Participants with an Abnormal Vital Signs/Peripheral Capillary Oxygen Saturation (SpO2) Reading as a Measure of Safety and Tolerability | Up to 28 days
  Number of participants with abnormal vital signs (including body temperature, heart rate, respiratory rate, systolic blood pressure [SBP], diastolic blood pressure [DBP]), and SpO2 measurements will be reported.
Number of Participants with an Abnormal Electrocardiogram (ECG) Reading as a Measure of Safety and Tolerability | Up to 28 days
  Number of participants with abnormal twelve-lead ECG will be reported.
Number of Participants with Clinical Laboratory Abnormalities as a Measure of Safety and Tolerability | Up to 28 days
  Number of participants with clinical laboratory abnormalities (clinical laboratory tests include the following: hematology panel, serum chemistry panel, urinalysis, estimated glomerular filtration rate (GFR), urine pregnancy test (women only), and serum procalcitonin levels) will be reported.
Maximum Observed Plasma Concentration (Cmax) of JNJ-63549109 | Dose 1: 0.5 to 1 hour postdose, and 2 to 3 hours postdose; Dose 2: predose, and 3 to 6 hours postdose; Dose 3 and 10: predose
  The Cmax is the maximum observed plasma concentration of JNJ-63549109. JNJ-63549109 is the metabolite of lumicitabine.
Concentration at 12 Hours Postdose (C12h) of JNJ-63549109 | Days 1, 2, and 5/6: 12 hours postdose
  The C12h is the predicted concentration of JNJ-63549109 at 12 hours postdose.
Area Under the Plasma Concentration-Time Curve (AUC) of JNJ-63549109 | Dose 1: 0.5 to 1 hour postdose, and 2 to 3 hours postdose; Dose 2: predose, and 3 to 6 hours postdose; Dose 3 and 10: predose
  AUC is defined as area under plasma concentration-time curve.
Ordinal Scale | Day of last dose (Day 5 or Day 6)
  The ordinal scale will be used to assess participant's status and consists of 6 categories that are exhaustive, mutually exclusive, and ordered, where: 1) Death, 2) Admitted to intensive care unit (ICU), 3) Non-ICU hospitalization requiring supplemental oxygen, 4) Non-ICU hospitalization not requiring supplemental oxygen, 5) Not hospitalized, unable to resume normal activities, 6) Not hospitalized, resumption of normal activities.
Length of Hospital Stay from Admission to Discharge | From admission to discharge (Up to 28 days)
  The length of hospital stay from admission to discharge will be reported.
Length of Hospital Stay from Admission to Readiness for Discharge | From admission to readiness for discharge discharge (Up to 28 days)
  The length of hospital stay from admission to readiness for discharge will be reported.
Length of Hospital Stay from Study Treatment Initiation to Discharge | From study treatment initiation to discharge (Up to 28 days)
  The length of hospital stay from study treatment initiation to discharge will be reported.
Length of Hospital Stay from Study Treatment Initiation to Readiness for Discharge | From study treatment initiation to readiness for discharge (Up to 28 days)
  The length of hospital stay from study treatment initiation to readiness for discharge will be reported.
Percentage of Participants Requiring Admission to the Intensive Care Unit (ICU) | Up to 28 days
  The percentage of enrolled participants requiring admission to the ICU will be reported.
Duration of ICU Stay | Up to 28 days
  In the event that a participant requires admission to the ICU, the duration for how long the participant remained in the ICU will be measured.
Percentage of Participants Requiring Oxygen Supplementation/Noninvasive Mechanical Ventilation Support | Up to 28 days
  The percentage of enrolled participants requiring oxygen supplementation/noninvasive mechanical ventilation support (for example [eg], nasal cannula, face mask, continuous positive airway pressure, bilevel positive airway pressure) above pre-hMPV infection status will be reported.
Duration of Oxygen Supplementation/Noninvasive Mechanical Ventilation Support | Up to 28 days
  The duration of oxygen supplementation/noninvasive mechanical ventilation support (eg, nasal cannula, face mask, continuous positive airway pressure, bilevel positive airway pressure) above pre-hMPV infection status will be measured.
Percentage of Participants Requiring Invasive Mechanical Ventilation Support | Up to 28 days
  The percentage of enrolled participants requiring invasive mechanical ventilation support (eg, endotracheal-mechanical ventilation or mechanical ventilation via tracheostomy) above pre-hMPV infection status will be reported.
Duration of Invasive Mechanical Ventilation Support | Up to 28 days
  The duration of invasive mechanical ventilation support (eg, endotracheal-mechanical ventilation or mechanical ventilation via tracheostomy) above pre-hMPV infection status will be measured.
Time to no Longer Requiring Supplemental Oxygen | Up to 28 days
  The time to which a participant no longer requires supplemental oxygen will be measured.
Time to Clinical Stability | Up to 28 days
  Time to clinical stability is defined as the time at which the following criteria are all met: normalization of blood oxygen level (return to baseline; by pulse oximetry) without requirement of supplemental oxygen beyond baseline level, normalization of oral feeding, normalization of respiratory rate and normalization of heart rate.
Number of Hours from Initiation of Study Treatment Until SpO2 is Greater Than or equal to (>=) 93 Percent (%) on Room air | Up to 28 days
  The number of hours until SpO2 is >= 93% on room air among participants who were not on supplemental oxygen prior to onset of respiratory symptoms will be recorded.
Time for Respiratory Rate to Return to Pre-hMPV Infection Status | Up to 28 days
  The time for respiratory rate to return to pre-hMPV infection status will be recorded.
Time for Peripheral Capillary Oxygen Saturation (SpO2) Return to Pre-hMPV Infection Status | Up to 28 days
  The time for SpO2 to return to pre-hMPV infection status will be recorded.
Time for Body Temperature to Return to Pre-hMPV Infection Status | Up to 28 days
  The time for body temperature to return to pre-hMPV infection status will be recorded.
Percentage of Enrolled Participants Who Require Hydration and/or Feeding by Intravenous (IV) Catheter or Nasogastric Tube | Up to 28 days
  The percentage of enrolled participants who require hydration and/or feeding by intravenous (IV) catheter or nasogastric tube will be reported.
Number of Participants With Bacterial Superinfections Reported as AEs | Up to 28 days
  The number of participants with bacterial superinfections, as defined by the investigator based on clinical judgment and/or increasing procalcitonin levels, reported as AEs will be reported.
Number of Participants With Treatment-Emergent Complications | Up to 28 days
  The number of participants with treatment-emergent complications, including cardiovascular events and cerebrovascular events (for example, myocardial infarction, congestive heart failure exacerbation, arrhythmia, stroke) or Clostridium difficile-associated diarrhea, will be reported.
Change From Baseline in the National Early Warning Score (NEWS) Over Time | Baseline up to 28 days
  The NEWS scoring system measures acute-illness severity using 7 physiological parameters (respiration rate, oxygen saturation, supplementary oxygen requirement, temperature, systolic blood pressure, heart rate, and level of consciousness). Each parameter is scored between 0 and 3 compared to normal ranges, with higher scores indicating greater severity. The total score is the sum of the individual physiological parameter values and ranges between 0 (least severe) and 21 (most severe).
Number of Participants With All-Cause Mortality | Up to 28 days
  Number of participants will be assessed for all-cause mortality.
Time to Return to Pre-hMPV Infection Functional Status (Katz Activities of Daily Living [ADL] score) | Up to 28 Days
  Katz activities of daily living will assess questions related to Bathing, Dressing, Toileting, Transferring, Continence and Feeding. For the six individual activities, a score of 1 indicates independence, and a score of 0 indicates dependence. Total score will be calculated by adding the scores of all six activities and ranges from 0 high (participant independent) to 6 low (participant very dependent).
hMPV Viral Load Over Time | Up to 28 days
  Viral load over time will be measured in mid-turbinate nasal swabs (obtained from non-intubated participants) or in mid-turbinate nasal swabs and endotracheal samples (obtained from intubated participants or via suction through tracheostomy or other sampling methods) by qRT-PCR.
Peak hMPV Viral Load | Up to 28 days
  Peak viral load over time will be measured by qRT-PCR.
Time to Peak hMPV Viral Load | Up to 28 days
  Time to peak viral load as measured by qRT-PCR will be reported.
Rate of Decline of hMPV Viral Load | Up to 28 days
  Rate of decline in hMPV viral load during treatment as measured by qRT-PCR will be reported.
Time to hMPV Ribonucleic Acid (RNA) Being Undetectable | Up to 28 days
  Time to hMPV RNA being undetectable as measured by qRT-PCR.
Percentage of Participants With Undetectable hMPV Viral Load at Each Timepoint | From Day 1 to Day 7 and on Day 10, Day 14, and Day 28
  Percentage of participants with undetectable viral load at each time point will be reported.
AUC of hMPV Viral Load From Baseline up to Day 10 | Baseline up to Day 10
  The AUC of hMPV RNA log10 viral load (measured by qRT-PCR in the mid-turbinate nasal swab specimens) is estimated by analyzing mean log10 viral load values over time using a restricted maximum likelihood based repeated measures approach.
AUC of hMPV Viral Load from Baseline up to Day 14 | Baseline up to Day 14
  The AUC of hMPV RNA log10 viral load (measured by qRT-PCR in the mid-turbinate nasal swab specimens) is estimated by analyzing mean log10 viral load values over time using a restricted maximum likelihood based repeated measures approach.
AUC of hMPV Viral Load in Participants Assigned to a Longer Dosing Duration From Baseline Until 1 day After the Last Dose of Study Drug | Baseline Until 1 day After the Last Dose of Study Drug (approximately up to 12 days)
  If dosing duration is increased by the Independent Data Monitoring Committee (IDMC), the AUC of hMPV viral load (measured by qRT-PCR in the mid-turbinate nasal swab specimens) will be estimated by analyzing mean log10 viral load values over time using a restricted maximum likelihood based repeated measures approach.
Number of Participants With Postbaseline Changes in the hMPV Polymerase Lgene and Other Regions of the hMPV Genome Compared With Baseline Sequences | Up to 28 days
  Number of participants will be assessed for postbaseline changes in the hMPV polymerase Lgene (only if no mutations are seen in the Lgene) and other regions of the hMPV genome compared with baseline sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (112):
- United States (7):
  - UCSF Fresno, Fresno, California
  - MemorialCare Research Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Lake Internal Medicine Associates, Eustis, Florida
  - Northwestern University - Northwestern Memorial Hospital - Infectious Disease Center, Chicago, Illinois
  - St Michaels Medical Center, Newark, New Jersey
  - SUNY Upstate Medical University, Syracuse, New York
  - Marshfield Clinic, Marshfield, Wisconsin
- Argentina (8):
  - Hospital Regional Español, Bahía Blanca
  - Hospital Interzonal General de Agudos Dr. Jose Penna, Bahía Blanca
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - CEMIC Saavedra, Ciudad de Buenos Aires
  - Hospital Italiano de La Plata, Ciudad de La Plata
  - Hospital Rawson, Córdoba
  - Hospital Privado-Universitario de Cordoba, Córdoba
  - Instituto Medico Platense, La Plata
- Australia (7):
  - Queen Elizabeth Hospital, Adelaide
  - Flinders Medical Centre, Adelaide
  - Princess Alexandra Hospital, Brisbane
  - Barwon Health - University Hospital Geelong, Geelong
  - Royal Melbourne Hospital, Melbourne
  - Mater Hospital Brisbane, South Brisbane
  - Westmead Hospital, Sydney
- Brazil (5):
  - Hospital São Lucas da Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto
  - Hospital Sirio Libanes, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da Universidade De Sao Paulo, São Paulo
- Bulgaria (4):
  - MHAT 'Sv. Ivan Rilski' Kozloduy EOOD, Kozloduy
  - Specialized Hospital for Active Treatment of Pulmonary Diseases - Pernik, Pernik
  - Specialized Hospital for Active Treatment of Pulmonary Diseases - Troyan EOOD, Troyan Municipality
  - MHAT Dr Stefan Cherkezov, Veliko Tarnovo
- France (13):
  - CHU Rouen, Bois-Guillaume
  - CHU caen, Caen
  - Hôpital Louis Mourier, Colombes
  - APHP - Hopital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CHU Grenoble, La Tronche
  - CHU Nîmes, Nîmes
  - Hopital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - CHU la milétrie, Poitiers
  - CHU Saint-etienne, Saint-Priest-en-Jarez
  - Hopital Foch, Suresnes
  - Centre Hospitalier Universitaire de Tours, Tours
- Japan (20):
  - Fukuoka University Hospital, Fukuoka
  - National Hospital Organization Ibarakihigashi, Funaishikawa
  - Ogaki Municipal Hospital, Gifu
  - National Hospital Organization Tenryu Hospital, Hamamatue
  - Japanese Red Cross Nagasaki Genbaku Isahaya Hospital, Isahaya
  - Shimane University Hospital, Izumo
  - Shinkomonji hospital, Kitakyushu
  - Kobe City Medical Center General Hospital, Kobe
  - Japanese Red Cross Society Nagano Hospital, Nagano
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Higashinagoya National Hospital, Nagoya
  - Rinku General Medical Center, Osaka
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ōta-ku
  - Tohoku Medical And Pharmaceutical University Hospital, Sendai
  - Saka General Hospital, Shiogama
  - National Hospital Organization Tokyo National Hospital, Tokyo
  - Okinawa Prefectural Chubu Hospital, Uruma
  - Okitama Public General Hospital, Yamagata
  - Shimonoseki City Hospital, Yamaguchi
  - Shin Yukuhashi Hospital, Yukuhashi
- Malaysia (7):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Pulau Pinang, George Town
  - Hospital Raja Perempuan Zainab Ii, Kota Bharu
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Hospital Miri, Miri
  - Hospital Taiping, Taiping
- Netherlands (3):
  - UMCG, Groningen
  - UMC Utrecht, Utrecht
  - Gelre Ziekenhuizen Zutphen, Zutphen
- Poland (5):
  - 10 Wojskowy Szpital Kliniczny z Poliklinika, Bydgoszcz
  - Wojewódzki Szpital Specjalistyczny im. św. Rafała w Czerwonej Górze, Chęciny
  - SSZZOZ im. dr Teodora Dunina w Rudce, Mrozy
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc w Olsztynie, Olsztyn
  - Samodzielny Publiczny Zespół Opieki Zdrowotnej w Proszowicach, Proszowice
- Russia (8):
  - State Health Care Institution 'Engels city hospital #2', Engel's
  - Saint-Petersburg State Health Care Institution 'Vvedenskaya Hospital', Saint Petersburg
  - Clinical Infectious Diseases Hospital n. a. S.P. Botkin, Saint Petersburg
  - Saint-Petersburg State Public Health Organization City Clinical Hospital #26, Saint Petersburg
  - Regional State Health Care Institution 'Clinical Hospital #1', Smolensk
  - Siberian State Medical University, Tomsk
  - State Health Care Institution of Voronezh region 'Voronezh regional clinical infectious hospital', Voronezh
  - Clinical Emergency Hospital n.a. N.V. Solovyev, Yaroslavl
- South Korea (6):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Yeungnam University Medical Center, Daegu
  - Gachon University Gil Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - Hosp. Gral. Univ. de Elche, Elche
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Alvaro Cunqueiro, Vigo
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skanes universitetssjukhus, Malmo
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (5):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taipei Municipal Wanfang Hospital, Taipei
- Ukraine (4):
  - Bukovian State Medical University, Dept. of Infectious Disease and Epidemiology, Chernivtsi
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Kharkiv National Medical University, Regional Clinical Infectious Hospital, Kharkiv
  - Vinnytsia City Clinical Hospital #1, Department of Infectious Diseases #1, Vinnytsia